CLINICAL TRIAL: NCT03816904
Title: Involvement of SK3 Calcium Channel in Taxane Neuropathy
Acronym: NEUROTAX
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18/NEUROTAX; 2018-A02884-51 (Other: IdRCB)
Record Dates: First submitted 2019-01-10; First posted 2019-01-25 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Chemotherapy-induced Peripheral Neuropathy; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — assay number of CAG triplets composing the KCNN3 gene usual blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast or prostate cancer: Taken blood samples on patients hospitalized in medical oncology day hospital at the University Hospital of Tours or CHC oncology day hospital, for their chemotherapy with taxanes (paclitaxel or docetaxel) for breast or prostate cancer
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples before the introduction of chemotherapy

SUMMARY:
Taxane neuropathy is a common and long-term side effect of long-term morbidity in patients surviving cancer. No preventive or symptomatic treatment has been shown to be effective. Its pathophysiology is poorly known and probably multifactorial. A possible mechanism would be mediated by the activation of the SK3 calcium channel: a retrospective study carried out at the University Hospital of Tours (Carina RUA) found a significant association between the number of CAG triplets in the KCNN3 gene coding for the SK3 channel and the appearance of a taxane neuropathy.

DETAILED DESCRIPTION:
Patients hospitalized in medical oncology day hospital at the University Hospital of Tours or CHC oncology day hospital, for their chemotherapy with taxanes (paclitaxel or docetaxel) for breast or prostate cancer, will be offered the study.

The mode of administration of chemotherapy and the usual follow-up will not be modified by the protocol The determination of the SK3 status will be made from an additional tube collected during a collection as part of the treatment at the first arrival in a day hospital (no more blood tests). Blood sample of 7mL. Shipments and analyzes of samples in Tours in the pharmacogenetics laboratory under the responsibility of Dr. BARIN-LE GUELLEC.

This study is non-invasive, without impact on the therapeutic management. The result of the polymorphism of SK3 will not be indicated in the record, so as not to influence the follow-up of the treatment and to allow an evaluation of the occurrence of peripheral neuropathy in blindness of the number of repetitions of the CAG triplet of the KCNN3 gene.

ELIGIBILITY:
Inclusion Criteria:

Breast Group

* Age ≥ 18 years
* Breast cancer
* Chemotherapy with paclitaxel or docetaxel
* Adjuvant or neoadjuvant chemotherapy in localized cancer or first-line treatment in metastatic cancer
* Signed informed consent

Prostate Group

* Age ≥ 18 years
* Metastatic prostate cancer
* Chemotherapy with docetaxel in 1st line
* Signed informed consent

Exclusion Criteria:

* Anteriority or concomitance of another chemotherapy provider of neuropathy (platinum salts)
* Another possible cause of neuropathy: diabetes, alcoholism, vitamin B9 / B12 deficiency, neurodegenerative disease, Raynaud's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in oncology day hospital for their chemotherapy with taxanes (paclitaxel or docetaxel) for breast or prostate cancer, will be offered the study.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Appearance of a neuropathy secondary to taxanes using Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) | From baseline and up to 4 months of follow-up
  Evaluation of neuropathy will be performed using non-invasive test, gold standard, Cancer Institute Common Terminology Criteria for Adverse Events
  Grading (from best to worst) :
  0 = normal
  1. = slight paresthesia, mild weakness (subjective)
  2. = moderate paresthesia, moderate weakness (objective)
  3. = severe paresthesia with functional disability, severe weakness
  4. = paralysis
Appearance of a neuropathy secondary to taxanes using Total neuropathy score clinical (TNSc) | From baseline and up to 4 months of follow-up
  Evaluation of neuropathy will be performed using non-invasive test, Total neuropathy score clinical
  Grading (from best to worst) :
  Sensory symptoms : 0 = none (N), 1 = symptoms limited finger or toes, 2 = Symptoms extend to ankle or wrist, 3 = Symptoms extend to knee or elbow, 4 = Symptoms above knees or elbow or functionally disabling Motor symptoms : 0 = N, 1 = slight difficulty, 2 = moderate difficulty, 3 = require help/assistance, 4 = paralysis Autonomic symptoms : 0 = N, 1 , 2, 3, 4 (number of symptoms) Pin sensibility and vibration sensibility : 0 = normal (n), 1 = reduced in fingers/toes, 2 = reduced to wrist/ankle, 3 = reduced to elbow/knee, 4 = reduced to above elbow/knee Strength : 0 = n, 1 = mild weakness, 2 = moderate weakness, 3 = severe weakness, 4 = paralysis Deep tendon reflexe : 0 = n, 1 = ankle reflex reduced, 2 = ankle reflex absent, 3 = ankle reflex absent, other reduced, 4 = all reflexes absent

SECONDARY OUTCOMES:
Occurence of adverses events to taxanes (dysgeusia, myalgia, digestive toxicity tearing, onycholysis.) | From baseline and up to 4 months of follow-up
  Each adverse event will be evaluated using CTCAE score grading (from best to worst) :
  * 0 : none
  * 1 : minimal
  * 2 : moderate
  * 3 : severe
  * 4 : very severe

CONTACTS AND LOCATIONS:
Overall Officials: Catherine BARBE, MD, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Department of Oncology, Hospital, Chinon, Chinon
  - Department of Medical Oncology, University Hospital, Tours, Tours